CLINICAL TRIAL: NCT04172454
Title: A Multicenter, Open-label,Phase 1b/2 Study for Safety and Efficacy of AK104, a PD-1/CTLA-4 Bispecific Antibody, in Selected Advanced Solid Tumors
Brief Title: Safety and Efficacy of AK104, a PD-1/CTLA-4 Bispecific Antibody, in Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-202
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumors; Melanoma
Keywords: Bispecific; PD1/CTLA4; PD-1/PD-L1 relapsed/refractory tumors
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 (Experimental): AK104 in subjects with advanced melanoma and other selected advanced solid tumor including PD-1/PD-L1 relapsed/refractory tumors)
  Interventions: Biological: AK104

INTERVENTIONS:
Biological: AK104 — AK104, 6mg/kg, Q2W

SUMMARY:
A multicenter, open-label, phase 1b/2 study to evaluate the safety and efficacy of AK104, a PD-1 and CTLA-4 bispecific antibody, in selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Male or female, age ≥ 18 years and ≤75, at the time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
4. Estimated life expectancy of ≥3 months.
5. Histologically or cytologically documented advanced or metastatic melanoma and other selected advanced solid tumors.
6. Subjects must have at least one measurable lesion per RECIST v1.1.
7. Available archived tumor tissue sample to allow for correlative biomarker studies. In the setting where archival material is unavailable or unsuitable for use , the subject must consent and undergo fresh tumor biopsy (biopsy at acceptable risk as judged by the investigator).
8. Adequate organ functions.
9. Female subjects of childbearing potential who are sexually active with a nonsterilized male partner must use an acceptable method of contraception from screening, and must agree to continue using such precautions for 90 days after the final dose of investigational product.
10. Subjects who agree to take effective contraception methods from screening to 120 days after the last dose of investigational product.
11. Willing to follow all the experimental requirements designated by the protocol.

Exclusion Criteria:

1. Prior use of investigational products or devices within 4 weeks prior to the first administration of the study treatment.
2. Concurrent enrollment into another clinical study, except the study belongs to investigational, non-interventional studies or the follow-up period of interventional studies.
3. Prior exposure to anti-tumor therapies, including systematic chemotherapy, radiotherapy, immunotherapy, hormone therapy, targeted therapy (within 2 weeks before the first administration of the study treatment), and systematic immune-modulators (including but not limited to interferon, interleukin-2 and tumor necrosis factor) within 4 weeks prior to the first administration of the study treatment. Prior exposure to Chinese herbal medicine or proprietary Chinese medicine with anti-tumor functions within 2 weeks prior to the first administration of the study treatment.
4. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria. Hair loss is excluded.
5. For subjects previously treated with anti-PD-1, PD-L1 or other immunotherapies: (1) Subjects have experienced a toxicity that led to permanent discontinuation of prior immunotherapy. (2) All AEs while receiving prior immunotherapy have not completely resolved or resolved to Grade 1 prior to screening for this study. (3) Subjects have required the use of additional immunosuppression other than corticosteroids for the management of an AE, or have experienced recurrence of an AE if re-challenged with corticosteroids while receiving prior immunotherapy.
6. Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with some exceptions.
7. Active or previously documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea).
8. Prior use of systematic corticosteroid (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to the first administration of the study treatment.
9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
10. Prior exposure to major surgery within 28 days prior to the first administration of the study treatment. Local procedures (eg, placement of a systemic port, core needle biopsy, and prostate biopsy) are allowed if completed at least 24 hours prior to the administration of the first dose of study treatment.
11. Known history of interstitial lung disease. The subjects highly suspected of interstitial lung disease will be excluded. Subjects with severe lung diseases affecting lung functions will be excluded.
12. Known history of active tuberculosis (TB). Subjects suspected of having active TB will be examined with x-ray, sputum, and clinical symptoms.
13. Known history of primary immunodeficiency virus infection or known history of testing positive for human immunodeficiency virus (HIV).
14. Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 1000 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
15. Serious infections within 4 weeks prior to the first dose of study drug.
16. Receipt of live, attenuated vaccination within 30 days prior to the first dose of study treatment, or plan to receive live, attenuated vaccine during the study.
17. Known history of sever hypersensitivity reaction to other monoclonal antibodies.
18. Known history of allergy or hypersensitivity to AK104 or any of its components
19. Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Anti-tumor activity of AK104 using objective response rate (ORR) based on RECIST v1.1 as assessed by the investigator | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Number of subjects experiencing adverse events (AEs) | From the time of informed consent through 90 days after last dose of AK104
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK104 until death due to any cause.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Minimum observed concentration (Cmin) of AK104 at steady state | From first dose of AK104 through to 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through to 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University; Xiaoshi Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Ma Y, Fan Y, Zhou J, Yang N, Yu Q, Zhuang W, Song W, Wang ZM, Li B, Xia Y, Zhao H, Zhang L. A multicenter, open-label phase Ib/II study of cadonilimab (anti PD-1 and CTLA-4 bispecific antibody) monotherapy in previously treated advanced non-small-cell lung cancer (AK104-202 study). Lung Cancer. 2023 Oct;184:107355. doi: 10.1016/j.lungcan.2023.107355. Epub 2023 Aug 29. PMID 37677918